CLINICAL TRIAL: NCT03461887
Title: Effects of a Long-term Home-based Exercise Training Program Using Minimal Equipment vs. Usual Care in COPD Patients: a Multicenter Randomized Controlled Trial
Brief Title: Home-based Exercise Training for COPD Patients
Acronym: HOMEX-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HOMEX-1
Record Dates: First submitted 2018-02-06; First posted 2018-03-12 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Chronic Disease; Lung Diseases, Obstructive; Respiratory Disease
Keywords: exercise; minimal equipment; home-based; COPD
MeSH Terms: conditions — Chronic Disease; Lung Diseases, Obstructive; Respiration Disorders; Motor Activity; Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): Home-based, minimal equipment exercise training program.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Usual care (study participation does not have any impact on regular treatment or treatment decisions, including participation in other exercise training programs or rehabilitation programs)

INTERVENTIONS:
Behavioral: Exercise — Home-based exercise training program that requires only minimal equipment, and is individually adaptable to the participant's exercise level (6 times per week; 15-20 min; 38 exercise cards and one interactive training agenda booklet). After randomization, a health care professional (HOMEX coach) will visit the intervention group participants at their home to set up the training location, to instruct the exercises and to establish individualized goals. Follow-up visits are planned after 3 and 8-9 weeks. Regular telephone calls will be conducted by the same HOMEX coach to motivate the patients, to discuss training progress and concrete benefits and barriers, and to adapt goals and the training program. Additional intervention elements are that a relative or friend is involved as a "sparring" partner to support the participant. The general practitioner is informed about the participation of his/her patient in the intervention.
  Arms: Exercise intervention

SUMMARY:
The aim of this study is to assess the effectiveness of a home-based exercise training program in COPD patients who have completed a pulmonary rehabilitation.

DETAILED DESCRIPTION:
Exercise training is an important component of the management of chronic obstructive pulmonary disease (COPD) and numerous trials have shown large improvements in health-related quality of life (HRQoL) and exercise capacity in persons with COPD. However, the great majority of patients who would benefit from pulmonary rehabilitation (PR) never follow such a program. Moreover, many COPD patients are either not instructed to exercise at all or fail to adhere to exercise training at home after completing pulmonary rehabilitation.

This study evaluates an exercise training program that requires minimal equipment (i.e., only a chair and elastic bands) and can be easily implemented long-term in the patient's home-setting.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent after being informed
* Diagnosis of COPD, defined as forced expiratory volume in 1s/forced vital capacity (FEV1/FVC)<70% predicted, FEV1<80 % predicted after bronchodilation, with or without chronic symptoms (cough, sputum production) corresponding to a GOLD stage II-IV
* Completion of an inpatient or outpatient pulmonary rehabilitation not longer than 1 months ago
* Male and female patients ≥40 years of age
* Knowledge of German language to understand study material and assessments

Exclusion Criteria:

* Patients not able to conduct the exercise training program due to physical, cognitive or safety reasons, as judged by investigator; e.g., lower limb joint surgery within preceding 3 months, unstable cardiac disease, predominant neurological limitations.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea | Change from baseline to 12 months
  Dyspnea domain of the Chronic Respiratory Questionnaire (CRQ); 5 questions; 7-point Likert-type scale ranging from 1 (most severe dyspnea) to 7 (no dyspnea)

SECONDARY OUTCOMES:
Dyspnea | Change from baseline to 3, 6 and 12 months
  Dyspnea domain of the Chronic Respiratory Questionnaire (CRQ); 5 questions; 7-point Likert-type scale ranging from 1 (most severe dyspnea) to 7 (no dyspnea)
Exercise capacity | Change from baseline to 12 months
  Six-Minute Walk Test (walk distance) and
  1-min Sit-to-Stand Test (number of repetitions)
Health-related quality of life | Change from baseline to 12 months
  Chronic Respiratory Questionnaires (CRQ): Fatigue, emotional function, mastery domain and EuroQoL (EQ-5D-5L): 5 Dimensions - Mobility, self-care, usual activities, pain/discomfort, anxiety/depression including 1 item each with 5 levels
Health status | Change from baseline to 12 months
  Visual analogue scale "Feeling thermometer" (0-100 scale; 0= "worst health you can imagine"; 100="best health you can imagine")
Exacerbations | During entire study, assessed at 12 months
  Event based, patient reported
Symptoms | Change from baseline to 12 months
  Questionnaire, COPD Assessment Test

OTHER OUTCOMES:
Compliance to the exercise training program | Assessed daily by intervention group participants during 12 months
  Percentage of fulfilled training sessions based on training diaries
Satisfaction with the exercise training program | From baseline to 12 months
  Questionnaire (Likert-Type scales)
Experience with the exercise training program | From baseline to 12 months (assessed at 12 months)
  Semi-structured interview
Health professionals' feedback | Assessed at 12 months
  Semi-structured interview
Cost effectiveness | From baseline to 12 months (assessed at 3, 6, 12 months)
  Questionnaire: cost per quality-adjusted life year

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - Klinik Barmelweid, Barmelweid
  - Berner Reha Zentrum AG, Heiligenschwendi
  - Zürcher RehaZentren Wald, Wald
  - Kantonsspital Winterthur, Winterthur
  - University of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Frei A, Radtke T, Dalla Lana K, Brun P, Sigrist T, Spielmanns M, Beyer S, Riegler TF, Busching G, Spielmanns S, Kunz R, Cerini T, Braun J, Tomonaga Y, Serra-Burriel M, Polhemus A, Puhan MA. Effectiveness of a Long-term Home-Based Exercise Training Program in Patients With COPD After Pulmonary Rehabilitation: A Multicenter Randomized Controlled Trial. Chest. 2022 Dec;162(6):1277-1286. doi: 10.1016/j.chest.2022.07.026. Epub 2022 Aug 8. PMID 35952766
- [Derived] Frei A, Radtke T, Dalla Lana K, Braun J, Muller RM, Puhan MA. Effects of a long-term home-based exercise training programme using minimal equipment vs. usual care in COPD patients: a study protocol for two multicentre randomised controlled trials (HOMEX-1 and HOMEX-2 trials). BMC Pulm Med. 2019 Mar 1;19(1):57. doi: 10.1186/s12890-019-0817-7. PMID 30823913